CLINICAL TRIAL: NCT01417260
Title: Effects of Breast Feeding on Post-Cesarean and Post-Vaginal Delivery Pain
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, Associate Professor, Stanford University
Other Study IDs: SU-08092011-8247; IRB 22053
Record Dates: First submitted 2011-08-11; First posted 2011-08-16 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Nocebo: Told breastfeeding may worsen pain
- No treatment: Told nothing
- Placebo: Told will improve pain

SUMMARY:
Oxytocin is a hormone that is released in response to distension of the cervix and uterus during labor, and after breast feeding as a result of nipple stimulation. In addition to oxytocin facilitating birth and breastfeeding, oxytocin has a number of effects on maternal behavior including bonding, social recognition, anxiolysis, sexual arousal.

The role of oxytocin in pain modulation has recently been highlighted. Intranasal or intrathecal (spinal) administration has been found to impact pain modulation. The administration of intravenous oxytocin has not provided effective analgesia because oxytocin is unable to pass to your brain. The role of breastfeeding on analgesia is poorly investigated, which is why we are carrying out this study.

DETAILED DESCRIPTION:
Patients will be recruited by a member of the research team when the patient is admitted to labor or delivery and when they are in the post-natal floor.

Patients will be divided into two groups initially depending on mode of delivery, vaginal vs. cesarean. The vaginal delivery group will be randomized into three groups. One group will be told that we are investigating the effect of oxytocin on pain intensity, the second group will be told that it reduces pain intensity, the third group will be told that it increases pain intensity.

The cesarean group are not going to be randomized, they will be told we are investigating the effect of oxytocin on pain intensity.

Demographic and obstetric will be collected by patient questioning as well as from the medical record on Day 1 post delivery. Analgesia data from the medical record will also be collected on days 1 and 2 post-delivery.

The primary outcome measure will be change in pain scores (0=no pain, 10=worse pain imaginable) during and after breastfeeding compared to pain before. We will examine both vaginal, cramping and surgical pain as appropriate.

The patients will be given a breastfeeding diary to complete, which will record the average pain scores (0-10) before, during and after each breastfeed.

Secondary outcome measure will include: Depression, PTDS, and other outcome measures. Patients will also be asked to complete pain intensity and depression (The Edinburgh Depression Scale) and a PTSD questionnaires. We will also determine pain preferences as relating to pain intensity and duration by another questionnaire.

At 6 weeks post-delivery, a member of the research team will call the participant to ask questions regarding current pain scores, success of breastfeeding and weight of the baby.

The study end-point is 6 weeks post-delivery. We will debrief participants who had deception at completion of the whole study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 40 yrs
2. ASA 1 or 2
3. Singleton gestation
4. Greater or equal to 37 weeks gestation
5. Vaginal delivery
6. Scheduled cesarean delivery with a Pfannenstiel incision

Exclusion Criteria:

1. Chronic pain
2. Patients prescribed regular analgesia medication ante-natally
3. Substance abuse
4. Classical cesarean incision
5. Emergency cesarean delivery
6. Patients not planning to breastfeed
7. Psychiatric or cognitive disorder, including anxiety or depression
8. Physicians, labor and delivery nurses, midwives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 30 patients posy cesarean delivery. 100 patients post vaginal delivery.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain in relation to breastfeeding | 6 weeks post-delivery
  The primary outcome measure will be change in pain scores (0=no pain, 10=worse pain imaginable) during and after breastfeeding compared to pain before. We will examine both vaginal, cramping and surgical pain as appropriate.
  The patients will be given a breastfeeding diary to complete, which will record the average pain scores (0-10) before, during and after each breastfeed.

SECONDARY OUTCOMES:
To determine the effects of suggestion and mood on pain | 6wks
  Secondary outcome measure will include: Depression, PTDS, and other outcome measures. Patients will also be asked to complete pain intensity and depression (The Edinburgh Depression Scale) and a PTSD questionnaires. We will determine the effects of suggestion (placebo vs. nocebo) on the pain experience.
  At 6 weeks post-delivery, a member of the research team will call the participant to ask questions regarding current pain scores, success of breastfeeding and weight of the baby.
  The study end-point is 6 weeks post-delivery.
To understand patients' preference for duration versus intensity of pain | 48 h
  We will also determine pain preferences as relating to pain intensity and duration by another questionnaire we have developed.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States